CLINICAL TRIAL: NCT00206661
Title: Phase 1/2 Safety, Pharmacokinetic, and Pharmacodynamic Study of Sargramostim (Leukine®) in Pediatric Patients With Active Crohn's Disease, With One-year Surveillance and Retreatment Extension
Brief Title: Safety and Efficacy Study in the Treatment of Pediatric Crohn's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 308001; 91409; Novel 6
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Crohn Disease
Keywords: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — sargramostim

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Sargramostim (Leukine)
- Arm 2 (Experimental)
  Interventions: Drug: Sargramostim (Leukine)

INTERVENTIONS:
Drug: Sargramostim (Leukine) — 4 mcg sargramostim with and without corticosteroids
  Other Names: BAY86-5326
  Arms: Arm 1
Drug: Sargramostim (Leukine) — 6 mcg sargramostim with and without corticosteroids
  Other Names: BAY86-5326
  Arms: Arm 2

SUMMARY:
The purpose of this study is to observe pediatric Crohn's Disease response to sargramostim in patients with or without steroid therapy at two possible dosage levels.

DETAILED DESCRIPTION:
On 29 May 2009, Bayer began transitioning the sponsorship of this trial to Genzyme. NOTE: This study was originally posted by sponsor Berlex, Inc. Berlex, Inc. was renamed to Bayer HealthCare, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Have a parent or guardian able to provide written informed consent
* Be able to provide verbal or written assent depending on age
* Age 6 to 16 years
* Have confirmed diagnosis of Crohn's Disease at study time of study entry based on radiologic, endoscopic, or histologic evaluations
* Have a PCDAI score >/= 30 points
* Have a negative serum pregnancy test within 7 days prior to receiving the first dose of sargramostim in female patients who, in the opinion of the investigator, are sexually active and of childbearing potential
* Be able to self-inject sargramostim or have a designee who can do so
* Available documentations of weight from 4 to 6 months prior to study entry

Exclusion Criteria:

* Existing colostomy or ileostomy
* Immediate need of GI surgery for active GI bleeding, peritonitis, intestinal obstruction, or intra-abdominal or perianal abscess requiring surgical drainage
* GI surgery within 3 month prior to receiving the first dose of sargramostim
* Symptoms of bowel obstruction or confirmed evidence of a clinically significant stricture within the last 6 month that has not been surgically corrected
* Use of any of the following medications within 4 weeks prior to receiving the first dose of study drug: 6 mercaptopurine, azathioprine, cyclophosphamide, methotrexate, mycophenolate mofetil, tacrolimus, cyclosporine, or thalidomide
* Use of licensed/registered and/or experimental anti-tumor necrosis factor (TNF) therapy such as infliximab or adalimumab within 8 weeks prior to first dose of sargramostim
* Use of any investigational drug within 4 weeks or 5 half-lives (whichever is greater) prior to receiving the first dose of sargramostim
* Concurrent use of corticosteroid therapy for Crohn's Disease, which exceeds a dose of 60 mg/day (or equivalent) of prednisone
* Inability to comply with protocol requirements or provide informed consent
* Presence of clinically important comorbid condition(s) unrelated to Crohn's Disease
* Prior use of recombinant human GM-CSF (sargramostim or molgramostim) or granulocyte colony-stimulating factor (G-CSF; filgrastim or pegfilgrastim)
* Current use of nutritional therapy (i.e., tube feeding or elemental/polymeric diet) which provides > 50% of daily caloric intake

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2004-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of sargramostim treatment with concomitant corticosteroid induction therapy | 12 weeks

SECONDARY OUTCOMES:
Characterize the pharmacokinetic, pharmacodynamics properties of sargramostim treatment with concomitant corticosteroid induction therapy | Week 0, 1, and 2
Evaluate the efficacy of sargramostim treatment with concomitant corticosteroids as measured by the Pediatric Crohn's Disease Activity Index (PCDAI), Physician's Global Assessment (PGA), and IMPACT-III Questionnaire | PCDAI, PGA: Week -1 to EOS; IMPACT-II: Week 0, 8 and EOS

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (7):
- United States (7):
  - San Francisco, California
  - Atlanta, Georgia
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Morristown, New Jersey
  - Philadelphia, Pennsylvania
  - Houston, Texas